CLINICAL TRIAL: NCT02965820
Title: Clinical Study of OPTI-FREE® PureMoist® for Presbyopic Contact Lens Wearers
Brief Title: OPTI-FREE® PureMoist® for Presbyopic Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: LCO115-P001
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Results first posted 2018-04-26 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-03

CONDITIONS: Presbyopia
Keywords: Contact lens induced dryness
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OFPM, then HMPS (Other): OPTI-FREE® PureMoist® multi-purpose contact lens solution in Period 1, followed by subject's habitual multi-purpose contact lens solution (HMPS) in Period 2. Each product used daily per packaging instructions with subject's habitual contact lenses for approximately 30 cleaning and disinfection cycles.
  Interventions: Device: Opti-Free® PureMoist® contact lens solution; Device: Habitual Multi-Purpose Contact Lens Solution; Device: Habitual Contact Lenses
- HMPS, then OFPM (Other): Subject's habitual multi-purpose contact lens solution in Period1, followed by OPTI-FREE® PureMoist® contact lens solution in Period 2. Each product used daily per packaging instructions with subject's habitual contact lenses for approximately 30 cleaning and disinfection cycles.
  Interventions: Device: Opti-Free® PureMoist® contact lens solution; Device: Habitual Multi-Purpose Contact Lens Solution; Device: Habitual Contact Lenses

INTERVENTIONS:
Device: Opti-Free® PureMoist® contact lens solution
  Other Names: OPTI-FREE® PureMoist®
Device: Habitual Multi-Purpose Contact Lens Solution
Device: Habitual Contact Lenses — Subject's habitual contact lens brand worn in a daily wear modality for 30 days.

SUMMARY:
The purpose of this study is to evaluate OPTI-FREE® PureMoist® (OFPM) compared to non-HYDRAGLYDE® multi-purpose contact lens solutions in presbyopes currently wearing soft contact lenses and experiencing symptoms of dryness.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent document;
* Current adapted two-week/monthly replacement soft contact lens wearers (at least 2 months) with symptoms of contact lens induced dryness;
* Near spectacle add of +0.50 or greater;
* Best corrected visual acuity (BCVA) to 20/30 or better in each eye at distance;
* Willing to wear lenses for a minimum of 5 days per week, 6 hours per day, and attend all study visits;
* Currently using a non-Alcon multi-purpose solution to care for lenses (at least 2 months);
* Use of digital devices (eg, smart phone, tablet, laptop computer, or desktop computer) for 20 consecutive minutes at least twice a week and willing to continue the same pattern for the duration of the study;
* Other protocol-specific inclusion criteria may apply.

Exclusion Criteria:

* Extended wear contact lens wearer (sleeps in lenses 1 or more nights per week);
* Any anterior segment infection, inflammation, disease, or abnormality that contraindicates contact lens wear as determined by the investigator;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the investigator, including use of any topical ocular medications that would require instillation during contact lens wear;
* Monocular (only 1 eye with functional vision) or fit with only 1 lens;
* Known sensitivity to any ingredients in OFPM;
* Prior refractive surgery;
* History of herpetic keratitis, ocular surgery, or irregular cornea;
* Pathological dry eye that precludes contact lens wear;
* Use of mechanical eyelid therapy or eyelid scrubs within 14 days before Visit 1 and not willing to discontinue during the study;
* Participation in any clinical study within 30 days of Visit 1;
* Currently using or have not discontinued Restasis®, Xiidra® or a topical steroid within the past 7 days;
* Other protocol-specific exclusion criteria may apply.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Manager, CPM, Study Director — Alcon, A Novartis Division

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 8 study centers located in the United States.
Pre-assignment Details: Of the 122 enrolled, 1 subject was exited as a screen failure prior to randomization. This reporting group includes all randomized subjects (121).
Groups:
- OFPM/HMPS: OPTI-FREE® PureMoist® (OFPM) multi-purpose contact lens solution in Period 1, followed by subject's habitual multi-purpose contact lens solution (HMPS) in Period 2. Each product used daily per packaging instructions with subject's habitual contact lenses for approximately 30 cleaning and disinfection cycles.
- HMPS/OFPM: Subject's habitual multi-purpose contact lens solution in Period1, followed by OPTI-FREE® PureMoist® contact lens solution in Period 2. Each product used daily per packaging instructions with subject's habitual contact lenses for approximately 30 cleaning and disinfection cycles.
Period: Period 1, First 30 Days
Arm/Group | OFPM/HMPS | HMPS/OFPM
Started | 59 | 62
Completed | 59 | 62
Not Completed | 0 | 0
Period: Period 2, Second 30 Days
Arm/Group | OFPM/HMPS | HMPS/OFPM
Started | 58 (One subject discontinued due to an AE after completion of Period 1 but before beginning Period 2.) | 62
Completed | 57 | 61
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects exposed to study lens care products (Full Analysis Set).
Groups:
- Overall: OFPM and HMPS used during Period 1 and Period 2 in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (5.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 119
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 101
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) Score at Day 30
Description: CLDEQ-8 score (assessment of contact lens discomfort) was obtained by adding the numerical responses to each of 8 items. Individual scales ranged from 0-4, 0-5, and 1-6, with a resultant overall score from 1 minimum to 37 maximum. A lower CLDEQ-8 score indicates less frequent or less intense symptoms.
Time Frame: Day 30, each product
Population: Full Analysis Set with non-missing responses
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- OFPM: OPTI-FREE® PureMoist® multi-purpose contact lens solution used daily per packaging instructions with subject's habitual contact lenses for approximately 30 cleaning and disinfection cycles.
- HMPS: Subject's habitual multi-purpose contact lens solution used daily per packaging instructions with subject's habitual contact lenses for approximately 30 cleaning and disinfection cycles.
Arm/Group | OFPM | HMPS
Number analyzed (Participants) | 120 | 119
units on a scale | 13.4 (7.42) | 15.8 (7.87)
Statistical Analysis 1: Comparison: OFPM vs HMPS; Test type: Superiority; p = 0.0030, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Day 1 through study completion, an average of 60 days
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational medical device. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator.
Groups:
- OFPM: All subjects exposed to OPTI-FREE® PureMoist® multi-purpose contact lens solution
- HMPS: All subjects exposed to habitual multi-purpose contact lens solution
Arm/Group | OFPM | HMPS
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/120
Serious Adverse Events (participants affected / at risk) | 1/121 | 0/120
Other Adverse Events (participants affected / at risk) | 0/121 | 0/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OFPM (N=121) | HMPS (N=120)
Knee operation (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2017-01-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT02965820/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT02965820/SAP_001.pdf